CLINICAL TRIAL: NCT04668586
Title: Laser Lithotripsy During Ureteroscopy - Holmium vs Thulium: A Clinical Prospective Randomized Trial of Effectiveness and Safety
Brief Title: Laser Lithotripsy During URS - Holmium vs Thulium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170907
Record Dates: First submitted 2020-12-06; First posted 2020-12-16 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Intervention Model Description: Arm 1: Holmium:YAG laser lithotripsy Arm 2: Thulium Fiber laser lithotripsy
Who Masked: Participant
Masking Description: The patient is in narcosis when the designated treatment is decided by randomisation, and the treatment is about to start.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Holmium:YAG laser machine (Experimental): The ureteral or renal stones planned for treatment with URS and laser lithotripsy are fragmented or dusted using a Holmium:YAG laser machine.
  Interventions: Device: Holmium:YAG laser machine
- Thulium Fiber laser machine (Experimental): The ureteral or renal stones planned for treatment with URS and laser lithotripsy are fragmented or dusted using a Thulium Fiber laser machine.
  Interventions: Device: Thulium Fiber laser machine

INTERVENTIONS:
Device: Holmium:YAG laser machine — Ureteroscopy with Holmium:YAG laser lithotripsy
  Arms: Holmium:YAG laser machine
Device: Thulium Fiber laser machine — Ureteroscopy with Thulium Fiber laser lithotripsy
  Arms: Thulium Fiber laser machine

SUMMARY:
The aim of the study is to compare URS lithotripsy performed with Holmium:YAG laser and Thulium Fiber Laser.

The study is designed as a prospective clinical randomised trial, where the study participants are randomised to either URS with Holmium:YAG laser or URS with Thulium Fiber Laser.

The outcomes of the URS procedures are compared for the two treatment arms.

DETAILED DESCRIPTION:
The primary aim of the study is to compare the stone free rate (SFR) following URS lithotripsy with Holmium and Thulium lasers. SFRs will be compared both for ureteral stones, renal stones and ureteral and renal stones in total.

Secondary aims are to compare the results of the two lasers in terms of operating times, intraoperative complications, postoperative complications and the rate of post endoscopic JJ-stenting.

The study is designed as a prospective clinical randomised trial, where the study participants are randomised to either URS with Holmium:YAG laser or URS with Thulium Fiber Laser.

The outcomes of the URS procedures are compared for the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for ureteroscopic treatment of ureteral and renal stones at the Day Surgery Unit at Haukeland University Hospital, Bergen, Norway

Exclusion Criteria:

* Known pathology of the upper urinary tract
* Untreated infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Ulvik, MD PhD, Principal Investigator — Helse-Bergen HF, Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No
IPF will not be available to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Holmium:YAG Laser Machine | Thulium Fiber Laser Machine
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Holmium:YAG Laser Machine | Thulium Fiber Laser Machine | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 54 [45 to 64] | 53 [38 to 68] | 53 [42 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 39 | 38 | 77
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Norway | 60 | 60 | 60
Stone size [Median (Inter-Quartile Range); unit: mm] — Population: Patients had either renal stones (n = 75) or ureteral stones (n = 45). The total number of participants were 120 (overall)
  mm
    Renal stones: number analyzed (Participants) | 39 | 36 | 75
    Renal stones | 12 [8 to 18] | 12 [7 to 16] | 12 [8 to 17]
    Ureteral stones: number analyzed (Participants) | 21 | 24 | 45
    Ureteral stones | 7 [6 to 10] | 8 [6 to 11] | 8 [6 to 10]
Stone location [Number; unit: participants] — Population: The total number of participants is 120. Some participants had stones in the renal pelvis (n=75) and some had stones in the ureter (n=45). The sum of participants with stones in the renal pelvis and ureter is 120.
  participants
    Renal stones - lower calyx: number analyzed (Participants) | 25 | 22 | 47
    Renal stones - lower calyx | 25 | 22 | 47
    Renal stones - all other locations: number analyzed (Participants) | 14 | 14 | 28
    Renal stones - all other locations | 14 | 14 | 28
    Ureteral stones - upper: number analyzed (Participants) | 11 | 6 | 17
    Ureteral stones - upper | 11 | 6 | 17
    Ureteral stones - middle: number analyzed (Participants) | 1 | 2 | 3
    Ureteral stones - middle | 1 | 2 | 3
    Ureteral stones - lower: number analyzed (Participants) | 9 | 16 | 25
    Ureteral stones - lower | 9 | 16 | 25

OUTCOME MEASURES:

1. Primary Outcome: Stone Free Rate
Description: Evaluation of stone free status on CT scan following URS. Stone free status is defined as no residual fragments.
Time Frame: 3 months after the URS
Measure: Count of Participants; unit: Participants
Arm/Group | Holmium:YAG Laser Machine | Thulium Fiber Laser Machine
Number analyzed (Participants) | 60 | 59
Participants | 34 | 47
Statistical Analysis 1: Comparison: Holmium:YAG Laser Machine vs Thulium Fiber Laser Machine; Test type: Superiority; p < 0.006, Chi-squared

2. Secondary Outcome: Operating Time
Description: Surgical operating time
Time Frame: Decided immediately after the surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Holmium:YAG Laser Machine | Thulium Fiber Laser Machine
Number analyzed (Participants) | 60 | 60
minutes | 60 [45 to 70] | 49 [32 to 63]
Statistical Analysis 1: Comparison: Holmium:YAG Laser Machine vs Thulium Fiber Laser Machine; Test type: Superiority; p = 0.008, t-test, 2 sided; Adjusted for four-category stratification group

3. Secondary Outcome: Intraoperative Complications
Description: Intraoperative complications leading to abruption of the URS procedure
Time Frame: Decided immediately after the surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Holmium:YAG Laser Machine | Thulium Fiber Laser Machine
Number analyzed (Participants) | 60 | 60
Participants | 0 | 0

4. Secondary Outcome: Postoperative Complications
Description: Postoperative complications (ie. infection, pain, stricture) leading to intervention or readmittance after the URS procedure.
Time Frame: Within 3 months post endoscopically
Measure: Count of Participants; unit: Participants
Arm/Group | Holmium:YAG Laser Machine | Thulium Fiber Laser Machine
Number analyzed (Participants) | 60 | 60
Participants
  Total participants needing readmission | 8 | 7
  Infection | 6 | 4
  Obstruction | 2 | 4
  Other | 1 | 1
Statistical Analysis 1: Comparison: Holmium:YAG Laser Machine vs Thulium Fiber Laser Machine; Test type: Superiority; p = 1, Chi-squared

5. Secondary Outcome: Postoperative JJ-stenting
Description: How many needed postendoscopic stunting following the URS procedure
Time Frame: Decided immediately after the surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Holmium:YAG Laser Machine | Thulium Fiber Laser Machine
Number analyzed (Participants) | 60 | 60
Participants | 31 | 22
Statistical Analysis 1: Comparison: Holmium:YAG Laser Machine vs Thulium Fiber Laser Machine; Test type: Superiority; p = 0.09, Chi-squared, Corrected; Adjusted for four-category stratification group

ADVERSE EVENTS:
Time Frame: From surgery until 3 months folloe-up
Description: Adverse events reported according to Clavien-Dindo classification
Arm/Group | Holmium:YAG Laser Machine | Thulium Fiber Laser Machine
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 8/60 | 7/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Holmium:YAG Laser Machine (N=60) | Thulium Fiber Laser Machine (N=60)
Postoperative complications (Renal and urinary disorders) | 8 (60) | 7 (60) — Adverse Events were monitored/assessed in such a manner that the specific Adverse Event Terms cannot be separated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT04668586/Prot_SAP_000.pdf